CLINICAL TRIAL: NCT03552068
Title: Study of Clonidine Efficacy for the Treatment of Impulse Control Disorders in Parkinson's Disease: A Pilot Double Blind Randomized Trial
Brief Title: Study of Clonidine Efficacy for the Treatment of Impulse Control Disorders in Parkinson's Disease:
Acronym: ID-CLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69HCL18_0135; 2019-000165-20 (EudraCT Number)
Record Dates: First submitted 2018-05-17; First posted 2018-06-11 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease; Mpulse Control Disorders
Keywords: Parkinson's disease; Impulse control disorder; Clonidine; Noradrenergic system
MeSH Terms: conditions — Parkinson Disease; Disruptive, Impulse Control, and Conduct Disorders | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients under placebo (Placebo Comparator): Treatment will be taken during 8 weeks with one visit at 2, 4 and 8 weeks. The usual antiparkinsonian treatment of the patient should remain stable throughout the 8 weeks.
  Interventions: Drug: placebo
- Patient under clonidine (Active Comparator): Treatment will be taken during 8 weeks with one visit at 2, 4 and 8 weeks. The usual antiparkinsonian treatment of the patient should remain stable throughout the 8 weeks.
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: placebo — Treatment (placebo) will be taken during 8 weeks with one visit at 2, 4 and 8 weeks.
  Medication: placebo twice a day (in the morning and evening).
  Arms: Patients under placebo
Drug: Clonidine — Treatment will be taken during 8 weeks with one visit at 2, 4 and 8 weeks. Medication: 75 μg of clonidine twice a day (in the morning and evening).
  Arms: Patient under clonidine

SUMMARY:
Noradrenergic system is involved in impulsivity in the general population and is altered in Parkinson's disease (PD) in the early stages of the disease. Thus, targeting this system could be of interest in impulse control disorder (ICD). Acting on the noradrenergic system is possible using clonidine, an α2 adrenergic agonist largely used in hypertension treatment and that induces a decrease of NADR release. Thus, our aim is to conduct a proof of concept study evaluating the efficacy and safety of clonidine on ICD in PD. This study is a multicenter, randomized, double-blind, placebo-controlled in parallel group clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PD according to MDS (movement disorders society) criteria for at least one year
* Patients with ICD with a QUIP-RS score ≥10 and/or at least one of the sub-scores in the following range: Pathological gambling between >6 and 12; Pathological gambling between >8 and 12; Hypersexuality between > 8 and 12; Eating between > 7 and 12. The use of "lower" margins will guarantee that patients will present behavioral disturbances severe enough to justify clonidine treatment. On the other hand, the use of "upper" margins will guarantee that the patients included in the trial will not suffer from ICD too severe to ethically participate to a placebo controlled study.
* Weight between 40 and 95kg
* Stable antiparkinsonian medication since at least 2 months before randomization and medication supposed to remain stable during the study
* ICD onset after Parkinson's disease onset and after initiation of dopaminergic drugs
* No signs of dementia (Montreal Cognitive Assessment, MOCA >20);
* No lactose intolerance which may compromise the tolerance of the placebo;
* Patients with health insurance
* Patients without judicial protection measure except directly linked to ICD
* For women of childbearing potential, an effective contraception method for at least 2 months before randomization (as implants or oral oestro-progestative contraceptives), condom use for men during the study. βHCG dosage in urine should be negative at randomization for women.

Exclusion Criteria:

Patients with major depression (BDI >19);

* Patients with another parkinsonian syndrome (Parkinson "plus" or vascular Parkinsonism)
* Orthostatic hypotension
* Patients with swallowing disorders that may prevent oral medication,
* Contraindication to clonidine: Hypersensibility; Severe bradyarythmia due to a cardiac disease
* Patients receiving a treatment potentially interacting with clonidine
* Patients with Raynaud's disease or obliterating thromboangiitis
* Patients With Heart failure or severe coronary artery disease
* Patients with a drug treatment having a potential interaction with clonidine (see list, appendix 2);
* Presence of renal failure (Cockcroft-Gault at inclusion visit<30 ml/min/1,73m2);
* Patients with a present or past history of addiction (apart ICD) or with a substance abuse (except Tabaco)
* Pregnant or lactating women
* Already participating in another biomedical research project

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
QUIP-RS (Questionnaire for Impulsive-Compulsive Disorders in Parkinson's disease - Rating Scale) | at 8 weeks
  Diminution of impulse control disorder severity on the initial more elevated sub-score of the QUIP-RS between the first visit and the eighth week under clonidine.
  Diminution of impulse control disorder severity on the initial more elevated sub-score of the QUIP-RS between the first visit and the eighth week under clonidine.
  Diminution of impulse control disorder severity on the initial more elevated sub-score of the QUIP-RS between the first visit and the eighth week under clonidine.

SECONDARY OUTCOMES:
MDS-UPDRS | at 4 and 8 weeks
  The Movement Disorder Society Unified Parkinson Disease Rating
STAI | at 4 and 8 weeks
  State-Trait Anxiety Index
BDI II | at 4 and 8 weeks
  Beck Depression Inventory II It is a self-administered questionnaire each of them using a four-point ordinal scoring system. For the summary index the scores were standardized from 1 to 40, so that higher scores indicate higher depression.
ECMP scores | at 4 and 8 weeks
  Behavior evaluation of Parkinson's patients It is a self-administered questionnaire each of them using a four-point ordinal scoring system. For the summary index the scores were standardized from 1 to 40, so that higher scores indicate higher depression.
QUIP-RS sub-scores | at 4 weeks
  Questionnaire for Impulsive-Compulsive Disorders in Parkinson's disease - Rating Scale Diminution of impulse control disorder severity on the initial more elevated sub-score of the QUIP-RS between the first visit and the fourth weeks under clonidine.
  It is a self-administered questionnaire. For the summary index the scores were standardized from 1 to 112, so that higher scores indicate higher Impulse control disorder. The sub score are standardized between 0 and 16.
QUIP-RS total score | at 4 and 8 weeks
  Evolution of QUIP-RS total score and sub-scores Diminution of impulse control disorder severity on total score of the QUIP-RS between the first visit, the fourth and the eighth weeks under clonidine.
  It is a self-administered questionnaire. For the summary index the scores were standardized from 1 to 112, so that higher scores indicate higher Impulse control disorder.
PDQ 39 scale (Parkinson Disease Quotation) | at 4 and 8 weeks
  It is a self-administered questionnaire comprised of 39 questions, each of them using a five-point ordinal scoring system, from which a single summary index can be calculated. For the summary index the scores were standardized from 0 to 100, so that higher scores indicate poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: LAURENCIN Chloé, Dr, Study Director — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laurencin C, Timestit N, Marques A, Duchez DD, Giordana C, Meoni S, Huddlestone M, Danaila T, Anheim M, Klinger H, Vidal T, Fatisson M, Caire C, Nourredine M, Boulinguez P, Dhelens C, Ballanger B, Prange S, Bin S, Thobois S. Efficacy and safety of clonidine for the treatment of impulse control disorder in Parkinson's disease: a multicenter, parallel, randomised, double-blind, Phase 2b Clinical trial. J Neurol. 2023 Oct;270(10):4851-4859. doi: 10.1007/s00415-023-11814-y. Epub 2023 Jun 20. PMID 37338615